CLINICAL TRIAL: NCT03374293
Title: Phase II Study of Radiation Therapy With Anti-PD-1 Antibody in Treating Patients With Unresectable Pancreatic Cancer
Brief Title: Combination of Radiation Therapy and Anti-PD-1 Antibody in Treating Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shixiu Wu (Other)
Responsible Party: Sponsor-Investigator, Shixiu Wu, director of the hospital, Hangzhou Cancer Hospital
Organization: Hangzhou Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH10
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; Radiation; Anti-PD-1 Antibody
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiation; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Radiation to 45-50.4 Gy, 5 x per week, 1.8Gy/fx. Radiation begun the day after the first dose of anti-PD-1 antibody . Anti-PD-1 antibody (every 2 weeks for 5 cycles) will be administered as an intravenous infusion over 30 minutes.
  Interventions: Radiation: Radiation; Drug: Anti-PD-1 Antibody

INTERVENTIONS:
Radiation: Radiation — RT to 45-50.4 Gy, 5 x per week, 1.8Gy/fx. Radiation begun the day after the first dose of anti-PD-1 antibody .
Drug: Anti-PD-1 Antibody — Anti-PD-1 antibody (every 2 weeks for 5 cycles) will be administered as an intravenous infusion over 30 minutes.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of radiation therapy combined with anti-PD-1 antibody in patients with pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or female.
2. Histologically or cytologically confirmed pancreatic cancer.
3. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
4. Can provide either a newly obtained or archival tumor tissue sample.
5. ECOG 0-1.
6. Life expectancy of greater than 12 weeks.
7. Adequate organ function.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Other malignancy within 5 years prior to entry into the study, expect for curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers.
3. Known central nervous system (CNS) metastases.
4. Subjects with any active autoimmune disease or history of autoimmune disease.
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. History of Interstitial Pneumonia or active non-infectious pneumonitis.
8. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C.
9. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent.
10. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy.
11. Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent.
12. Received a live vaccine within 4 weeks of the first dose of study medication.
13. Pregnancy or breast feeding. Decision of unsuitableness by principal investigator or physician-in-charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Local control | 2 year
  occurrence of local or regional progression

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 3 months
  Number of participants with treatment-related adverse events as assessed by Number of participants with treatment-related adverse events as assessed by treatment-related adverse events assessed by CTCAE v4.0
Objective response rate | 3 months
  Objective response rate as assessed by RECIST criteria
Overall survival | 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided